CLINICAL TRIAL: NCT04811586
Title: Efficacy and Safety of One-Step Hybrid Coronary Revascularization Versus Percutaneous Coronary Intervention for Patients With Multivessel Disease
Brief Title: Efficacy and Safety of One-Stage Hybrid Coronary Revascularization
Acronym: HCR-EAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCR-EAST
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: hybrid coronary revascularization (HCR); percutaneous coronary intervention (PCI); coronary artery bypass graft (CABG); multivessel coronary artery disease
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-step Hybrid Coronary Revascularization (HCR) (Experimental): One-step HCR is defined as off-pump MIDCAB LIMA-LAD revascularization immediately followed by PCI for at-least one non-LAD lesion(or LAD-diagonal lesion) with DES implantation in a hybrid operating room.
  Interventions: Procedure: coronary revascularization
- Percutaneous Coronary Intervention (PCI) (Active Comparator): PCI will be performed using standard technique at the discretion of interventional cardiologist with DES implantation in a routine catheter lab.
  Interventions: Procedure: coronary revascularization

INTERVENTIONS:
Procedure: coronary revascularization — to improve the blood supply for coronary arteries by using either percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)

SUMMARY:
Coronary revascularization could be accomplished either by percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG). PCI with drug-eluting stent (DES) implantation is featured by minimal invasive, low complication and rapid rehabilitation. CABG is characterized by improved long-term, event-free survival attributable to the use of left internal mammary artery (LIMA) graft. Hybrid coronary revascularization (HCR) consists of LIMA bypass to left anterior coronary descending artery (LAD) by minimal invasive direct coronary artery bypass (MIDCAB) and PCI of other stenosed coronary arteries with DES implantation. One-step HCR entails LIMA-LAD anastomosis performed through MIDCAB, immediately followed by PCI for non-LAD lesions, sometimes for diagonal branch, in the hybrid operating room. Limited data are available in comparing one-step HCR to PCI alone for the treatment of multivessel coronary artery disease(MVD). The current EAST-HCR study will investigate the efficacy and safety of one-step HCR for patients with MVD, as comparing to PCI alone.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years and older
2. signed the informed consent
3. indicated for revascularization, with possible bypass segment in LAD and amendable lesions by PCI in other vessels
4. anatomy requiring as following: (1) Multivessel CAD involving the LAD (proximal or mid) and/or LM (ostial, mid-shaft or distal) with at least 1 other epicardial coronary artery requiring treatment in LCX or RCA, including: (2) LAD disease, and a major diagonal lesion, either bifurcation or independent in location, with both requiring revascularization (determined by QFR or FFR) (3) LM distal bifurcation lesion (Medina 1,1,1), intended for 2-stent approach if randomized to PCI
5. Heart team discussion after angiogram, with conclusion of suitable candidate for either PCI or HCR
6. Able to tolerate and no plans to interrupt dual anti-platelet therapy for 3~12 months
7. Willing to comply with 2-year clinical follow-up

Exclusion Criteria:

1. Previous cardiac or thoracic surgery
2. Previous PCI of the LM and/or LAD within 12 months
3. Totally occluded left main vessel
4. Cardiogenic shock or LVEF <30%
5. Previous STEMI within 30-day prior to randomization
6. Concomitant vascular or other cardiac disease with plan of surgical treatment
7. Indication for chronic oral anticoagulation therapy
8. Previous stroke history within 6-month prior to randomization
9. Survival expectation less than 3 years due to non-cardiac illness
10. Allergy or hypersensitivity to any of the study drugs or devices used in the trial
11. Enrolled in additional clinical study
12. Informed consent not available or noncompliance with follow-up
13. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 2 years
  the occurrence of MACCE at 2 years' clinical follow-up, including all-cause death, myocardial infarction, stroke, and repeated revascularization

SECONDARY OUTCOMES:
Bleeding events | 2 years
  individual component of MACCE
Hospital duration (day) | up yo 2 years
Rate of complete revascularization at index hospitalization | 2 years
  rate of complete revascularization at index hospitalization (defined by Quantitative flow ration[QFR] or Fraction flow reserve[FFR])
Stent thrombosis event | 2 years
  stent thrombosis defined by Academic Research Consortium (ARC)

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhang, MD, PhD, Study Director — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China